CLINICAL TRIAL: NCT04790435
Title: Acute-On-Chronic Liver Failure In Cirrhotic Patients In Sohag University Hospital
Brief Title: Acute-On-Chronic Liver Failure In Cirrhotic Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eman Khalifa Al Sayed, Resident in Tropical Medicine and Gastroenterology Department, Sohag University
Other Study IDs: Soh-Med-21-02-12
Record Dates: First submitted 2021-03-01; First posted 2021-03-10 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Cirrhosis, Liver
Keywords: Cirrhosis, liver failure
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Liver Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cirrhosis is a condition characterized by diffuse fibrosis, severe disruption of the intrahepatic arterial and venous flow, portal hypertension and, ultimately, liver cell failure. Traditionally, cirrhosis has been dichotomised in compensated and decompensated, and the transition to decompensated cirrhosis happens when any of the following hallmarks occurs: presence of ascites, variceal haemorrhage and/ or hepatic encephalopathy (HE) . In Egypt, HCV is the main cause of liver cirrhosis followed by HBV

DETAILED DESCRIPTION:
Cirrhosis is a condition characterized by diffuse fibrosis, severe disruption of the intrahepatic arterial and venous flow, portal hypertension and, ultimately, liver cell failure. Traditionally, cirrhosis has been dichotomised in compensated and decompensated, and the transition to decompensated cirrhosis happens when any of the following hallmarks occurs: presence of ascites, variceal haemorrhage and/ or hepatic encephalopathy (HE). In Egypt, HCV is the main cause of liver cirrhosis followed by HBV. Once cirrhosis transitions from the compensated to the decompensated stage, it is associated with short-term survival (3-5 years) . The concept of acute-on-chronic liver failure (ACLF) has been widely used to study patients who underwent artificial support therapies as a bridge to liver transplantation (LT). In 2009, the Asian Pacific Association for the Study of the Liver (APASL) provided the first consensus on ACLF, defined as "an acute hepatic insult manifesting as jaundice and coagulopathy, complicated within 4 weeks by ascites and/or encephalopathy". In 2014, the definition was further expanded to include 'high 28-day mortality'. Therefore, acute on top of chronic liver failure (ACLF) is defined as a syndrome characterized by acute decompensated cirrhosis associated with failure of various organs and high short term mortality rate; based on CANONIC study which is a large scale prospective study, in which the kidneys were the most common affected organs, followed by liver, coagulation, the brain, circulation and the lungs. ACLF can occur in patients with chronic liver disease without cirrhosis (type A), with compensated cirrhosis (type B), and with decompensated cirrhosis (type C) .In many cases, a precipitating factor linked to the development of ACLF can be identified including alcohol intake, reactivation of HBV or acute hepatitis due to HAV or HEV, bacterial infection or GI hemorrhage. The CLIF-C OF score which consists of numbers and types of organ failures (OFs) including kidneys, liver, coagulation, the brain, circulation, and the lungs is associated with 28-day and 90-day mortality. Moreover, some specific organ dysfunction such as kidney dysfunction and moderate HE, when associated with single OF, was also associated with bad prognosis . On this background, diagnostic criteria of ACLF were established according to the presence, type and number of OFs.

The severity of ACLF was graded into different stages according to the number of OFs on ACLF grade 1, grade 2 and grade 3 and mortality correlates with ACLF severity.

To predict prognosis and mortality more accurately. developed CLIF-C-ACLF score which has a greater prognostic capability than CLIF-C- OF, It consists of the CLIF-C- OF combined with age and WBCs count. Few studies have addressed the patterns of acute on chronic liver failure in Egyptian cirrhotic patients . Therefore, we will conduct our study to shed

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients whether compensated or decompensated with an acute decompensation of cirrhosis which is defined by the recent development of ascites, encephalopathy, GI haemorrhage, bacterial infection, or any combination of these

Exclusion Criteria:

* no exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients whether compensated or decompensated with an acute decompensation of cirrhosis which is defined by the recent development of ascites, encephalopathy, GI haemorrhage, bacterial infection, or any combination of these
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Predictors of 28 day mortality rate in acute on chronic liver failure patients. with acute on top of chronic liver failure | 4 weeks from start point.
  It will be determined by univariate and multivariate analysis.

SECONDARY OUTCOMES:
Triggers of development of ACLF . | 4 weeks from start point.
  Alcohol intake, reactivation of HBV, acute hepatitis, bacterial infection, and GI haemorrhage
Types and numbers of organ failures in patients with ACLF. | 4 weeks from start point
  Kidneys, liver, coagulation, the brain, circulation, and the lungs.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
not decided